CLINICAL TRIAL: NCT05684666
Title: Effect of Slow Breathing and Progressive Muscle Relaxation Technique in Individual With Essential Hypertension: a Randomized Controlled Trial
Brief Title: Effect of Breathing and Muscle Relaxation Technique in Individual With Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Prinicipal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-07
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Autogenic Training; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SBE Group (Experimental): Slow Breathing Exercise (SBE) was performed by the participants of SBE group. Sixteen participants included in this group.
  Interventions: Other: Slow Breathing Exercise (SBE)
- PMR Group (Experimental): Progressive Muscle Relaxation (PMR) Technique was performed by the participants of the PMR group. It included 16-participants for the study.
  Interventions: Other: Progressive Muscle Relaxation (PMR) Technique
- Combined Group (Experimental): Sixty participants from the combined group performed both Slow Breathing Exercise and Progressive Muscle Relaxation technique in this study.
  Interventions: Other: Slow Breathing Exercise (SBE); Other: Progressive Muscle Relaxation (PMR) Technique
- Control Group (No Intervention): No intervention was received/performed by the sixteen participants of the control group in this study.

INTERVENTIONS:
Other: Slow Breathing Exercise (SBE) — Slow Breathing Exercise (SBE) delivered in a relaxed supine posture on a couch with keeping the feel flat and knee flexed to 90 degree.
  Participants were instructed to make six breaths per minute for 30 minutes per session, twice a week for 4 weeks.
  Arms: Combined Group; SBE Group
Other: Progressive Muscle Relaxation (PMR) Technique — Progressive Muscle Relaxation (PMR) Technique delivered in a relaxed supine posture on a couch with keeping the feel flat and knee flexed to 90 degree.
  Participants were instructed to complete all sixteen steps of PMR technique for 30 minutes per session, twice a week for 4 weeks.
  Arms: Combined Group; PMR Group

SUMMARY:
Primary hypertension, also called essential hypertension, is a rise in blood pressure (BP) with no identifiable cause. The most prevalent form of hypertension is essential hypertension, which involves 95% of patients with hypertension.Progressive muscle relaxation (PMR) is learning to relax some groups of muscles while paying attention to the feelings connected with both the tense and relaxed states.It is generally established that regular slow (deep) breathing exercises enhance respiratory and cardiovascular function by enhancing parasympathetic tone and reducing sympathetic activity, thus reducing BP, heart rate, respiratory rate, and stress levels in hypertensive patients. This study aimed to investigate the combined effect of slow breathing and PMR technique on BP, heart rate, respiratory rate, and anxiety in patients diagnosed with essential hypertension.

DETAILED DESCRIPTION:
From the previously published literature, it is obvious that both slow breathing and PMR and slow breathing is effective in patients with essential hypertension. However, no studies are available on the combined effect of these two techniques. So, the study aims to investigate the combined effect of slow breathing and PMR technique on BP, heart rate, respiratory rate, and anxiety in patients diagnosed with essential hypertension.

Sixty-four participants diagnosed with essential hypertension were randomly allocated into four groups (Slow breathing (SB), PMR, SB+PMR, Control) with 16 subjects in each. Baseline BP, HR, RR and perceived stress scale were taken. All three-intervention groups underwent 30 minutes of training three days before the day of the intervention. The intervention consisted of 30 minutes, pre, mid and post-intervention BP, HR, RR and Perceived Stress (PS) were measured. The control group rested for 30 minutes. Pre, mid and post-rest measurements of BP, HR, RR and PS were taken.

ELIGIBILITY:
Inclusion Criteria:

* Participants with essential hypertension, a diastolic BP between 90 to 109mm of Hg, a systolic BP of more than 140mm of Hg,
* Aged between 30 to 60 years, and
* Self co-operation.

Exclusion Criteria:

* Participants with secondary hypertension, any physical abnormalities that may disturb the exercise intervention,
* Participant who cannot perform any relaxation or breathing exercises, and
* Non-cooperation of participants.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | 8 Weeks
  SBP was measured using a portable electronic sphygmomanometer.
Diastolic Blood Pressure (DBP) | 8 Weeks
  DBP was measured using a portable electronic sphygmomanometer.
Heart Rate (HR) | 8 Weeks
  Heart Rate was measured using a portable electronic sphygmomanometer.
Respiratory Rate (RR) | 8 Weeks
  RR was measured manually as the number of breaths a participant takes per minute.
Perceived Stress (PS) | 8 Weeks
  Perceived Stress was assessed using the perceived stress scale (PSS) with ten items, each with a five-point Likert scale (where a score of 0 indicates "never," a score of 1 indicates "nearly never," a score of 2 "occasionally," a score of 3 "very often," and a score of 4 "often").

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Principal Investigator — King Saud University, Riyadh 11433, P.BOX 10219, Saudi Arabia
Locations (1):
- Rehabilitation Research Chair, Department of Rehabilitation Sciences, king Saud University, Riyadh, Riyadh 11433, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No